CLINICAL TRIAL: NCT05412446
Title: SPECT Imaging of Human Epidermal Growth Factor Receptor 2 (HER2) Expression in Primary Tumour and Metastatic Axillary Lymph Nodes Using Technetium-99m-labelled ADAPT6 Molecule-based 99mTc-ADAPT6.
Brief Title: 99mTc-ADAPT6 SPECT-based Non-invasive Quantification of HER2-expression in Breast Cancer With Metastatic Lymph Nodes
Acronym: 99mTc-ADAPT6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 99mTc-ADAPT6 in breast cancer
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Female
Keywords: 99mTc-ADAPT6; Breast Cancer; metastatic lymph nodes; HER2 expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Diagnostic Test: ADAPT6-SPECT Diagnostic SPECT for HER2 expression in primary tumour and metastatic lymph nodes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HER2-positive patients (Experimental): Maximum 15 evaluable subjects with HER2-positive status in primary tumour before chemo/targeted therapy have to be enrolled in the study.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: ADAPT6-SPECT
- HER2-negative patients (Experimental): Maximum 15 evaluable subjects with HER2-negative status in primary tumour before chemo/targeted therapy have to be enrolled in the study.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: ADAPT6-SPECT

INTERVENTIONS:
Drug: ADAPT6-SPECT — Diagnostic SPECT for HER2 expression in primary tumour and metastatic lymph nodes
  Other Names: Diagnostic ADAPT6-SPECT injection

SUMMARY:
An open-label, single center study with 99mTc-ADAPT6 SPECT and biopsies of primary tumour and metastatic lymph nodes in breast cancer patients, where the primary endpoint of the study is to find out the correlation between the HER2 expression measured by 99mTc-ADAPT6 SPECT and standard histopathology from relevant tumor and lymph node biopsies.

DETAILED DESCRIPTION:
Overall goal of the project: To determine HER2 expression level in primary breast cancer and axillary lymph node metastases before neoadjuvant targeted (trastuzumab or trastuzumab+pertuzumab) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Diagnosis of primary breast cancer with lymph node metastases
3. Availability of results from HER2 status previously determined on material from the primary tumor and metastatic LN, either a. HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive or b. HER2-negative, defined as a DAKO HercepTest™ score of 0 or 1+; or else if 2+ then FISH negative
4. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 109/L
   * Hemoglobin: > 80 g/L
   * Platelets: > 50.0 x 109/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
5. A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination

7. Subject is capable to undergo the diagnostic investigations to be performed in the study 8. Informed consent

Exclusion Criteria:

1. Any system therapy (chemo-/targeted therapy)
2. Second, non-breast malignancy
3. Active current autoimmune disease or history of autoimmune disease
4. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening) 4. Known HIV positive or chronically active hepatitis B or C
5. Administration of other investigational medicinal product within 30 days of screening
6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
SPECT/CT-based 99mTc-ADAPT6 uptake value in tumor lesions (SUV) | 2 hours
  SPECT/CT-based 99mTc-ADAPT6 uptake value in tumor lesions measured as 99mTc-ADAPT6 focal uptake coinciding with tumor lesions will be assessed using SPECT/CT at 2 hours after injection and measured in SUV
SPECT/CT-based 99mTc-ADAPT6 uptake value in metastatic lymph nodes (SUV) | 2 hours
  SPECT/CT-based 99mTc-ADAPT6 uptake value in metastatic lymph nodes SUV measured as 99mTc-ADAPT6 focal uptake coinciding with tumor lesions will be assessed using SPECT/CT at 2 hours after injection and measured in SUV
Tumor-to-background ratio (SPECT) | 2 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-ADAPT6 uptake coinciding with tumor lesions (SUV) will be divided by the value of 99mTc-ADAPT6 uptake coinciding with the regions without pathological findings (SUV)
LN-to-background LN ratio (SPECT) | 2 hours
  The SPECT-based LN-to-background LN ratio will be calculated as follows: the value of 99mTc-ADAPT6 uptake coinciding with LN lesions (SUV) will be divided by the value of 99mTc-ADAPT6 uptake coinciding with the regions without pathological findings (SUV)

SECONDARY OUTCOMES:
Matching test rate (percentage) | 2 hours
  Comparison of the 99mTc-ADAPT6 accumulation in the primary tumor and metastatic lymph nodes with the results of morphological and immunohistochemical studies.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD, PhD, Study Director — Caencer Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Tomsk NRMC, Tomsk, Russia